CLINICAL TRIAL: NCT01541306
Title: C-Type Natriuretic Peptide and Achondroplasia
Status: Completed | Type: Observational
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Alfred I. duPont Hospital for Children (Other); University of Otago (Other)
Responsible Party: Principal Investigator, Rob Olney, Physician/researcher, Nemours Children's Clinic
Other Study IDs: Nemours FL IRB 302926
Record Dates: First submitted 2012-02-13; First posted 2012-02-29 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Achondroplasia; Hypochondroplasia
Keywords: C-type natriuretic peptide; dwarfism; growth; achondroplasia; hypochondroplasia; biomarker
MeSH Terms: conditions — Achondroplasia; Hypochondroplasia; Dwarfism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum samples are stored for potential future research.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- achondroplasia or hypochondroplasia: Children or adults with achondroplasia or hypochondroplasia

SUMMARY:
Achondroplasia and hypochondroplasia are the most common forms of dwarfism. Recent studies have shown that a small hormone called C-type natriuretic peptide (CNP) is an important regulator of linear growth. The investigators believe that genetic abnormality that causes achondroplasia and hypochondroplasia also disrupts CNP signaling, which may contribute to the growth problem. The investigators propose to look at levels of this and other closely related hormones in children and adults with achondroplasia or hypochondroplasia to see if they are different from levels in healthy people. The investigators hypothesis is that CNP levels are elevated in children with achondroplasia or hypochondroplasia, compared the healthy population. Another hypothesis is that CNP levels are not elevated in adults with achondroplasia or hypochondroplasia, since adults have no growth-plate cartilage. By studying the potential role of the CNP system in achondroplasia and hypochondroplasia, not only will the investigators provide further insight into the pathophysiology of these common syndromes, the investigators will also provide greater insight into the regulation of normal linear growth.

DETAILED DESCRIPTION:
Achondroplasia is the most common form of dwarfism and is characterized by short limbs with the thighs and upper arms being the most affected. Achondroplasia is also associated with a narrowing of the foramen magnum and spinal stenosis. Hypochondroplasia is a related, but less severe form of dwarfism that does not have the neurologic problems. Achondroplasia and hypochondroplasia are caused by mutations in the fibroblast growth factor receptor-3 (FGFR-3) gene that causes constitutive activation of the receptor. FGFR-3 signals primarily through the MAP kinase pathway, which is overactivated in growth plate chondrocytes in achondroplasia. C-type natriuretic peptide (CNP) is a hormone that is produced and acts in the growth plate as a potent positive regulator of linear growth. CNP signals through natriuretic peptide receptor-B (NPR-B), generating cGMP. Studies in mice show that activation of the MAP kinase pathway inhibits signaling through NPR-B. Hence the achondroplasia phenotype may be due in part to inhibition of CNP signaling. Conversely, CNP intracellular signaling inhibits the MAP kinase pathway and CNP analogs are being studied as a potential specific therapy for achondroplasia. The objective of this project is to define the state of the CNP system in children and adults with achondroplasia or hypochondroplasia. Our hypotheses are 1) blood levels of CNP and its aminoterminal propeptide (NTproCNP) are elevated and blood levels of cGMP are reduced in children with achondroplasia or hypochondroplasia, due to inhibition of NPR-B; 2) CNP and NTproCNP levels are normal in adults with achondroplasia and hypochondroplasia, due to their lack of growth plate cartilage; and 3) as in healthy children, NTproCNP levels predict height velocity in children with achondroplasia or hypochondroplasia. These hypotheses will be addressed with two specific aims. Specific aim 1 is to determine plasma levels of CNP, NTproCNP, and cGMP in children and adults with achondroplasia or hypochondroplasia. Specific aim 2 is to determine if NTproCNP levels correlate with height velocity in children with achondroplasia or hypochondroplasia.

The study is an observational, cross-sectional/partially longitudinal study of children and adults with achondroplasia or hypochondroplasia. Children will be seen as part of routine clinic visits. Children seen more than once during the study period will provide longitudinal data. Adult subjects with achondroplasia or hypochondroplasia will be studied a single time. Data collected will include anthropometrics, information on neurologic complications of achondroplasia, and blood levels of CNP, NTproCNP, and cGMP. We anticipate 100 subjects will be recruited, with about 20 being studied as many as three times during the course of the study.

By studying the potential role of the CNP system in achondroplasia and hypochondroplasia, not only will we provide further insight into the pathophysiology of these common syndromes, we will also provide greater insight into the regulation of normal linear growth.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of achondroplasia or hypochondroplasia

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults with achondroplasia or hypochondroplasia
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
NTproCNP level in plasma | one time point
  Aminoterminal propeptide of CNP (NTproCNP) is measured in plasma by RIA and compared to an existing sex- and age- based reference range.

SECONDARY OUTCOMES:
CNP level in plasma | one time point
  C-type natriuretic peptide is measured in plasma by RIA and compared to an existing sex- and age- based reference range.
cGMP level in plasma | one time point
  Cyclic GMP levels are measured in plasma by RIA and compared to existing age- and sex- matched control samples.
Correlation between NTproCNP level and height velocity in children | Every six months over a period of a minumum of six months to a maximum of 2 years
  NTproCNP levels at baseline will be correlated with hieght velocity determined at subsequent visits. Measurements for determination of height velocity will be at least 6 months apart, but no more than 2 years apart. For subjects with multiple subsequent visits, the visit closest to 1 year after the baseline visit will be used for height velocity determination.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Olney, MD, Principal Investigator — Nemours Children's Clinic; Michael Bober, MD, PhD, Principal Investigator — Alfred I. duPont Hospital for Children
Locations (1):
- Alfred I. duPont Hospital for Children, Wilmington, Delaware, United States

REFERENCES:
- [Derived] Olney RC, Prickett TC, Espiner EA, Mackenzie WG, Duker AL, Ditro C, Zabel B, Hasegawa T, Kitoh H, Aylsworth AS, Bober MB. C-type natriuretic peptide plasma levels are elevated in subjects with achondroplasia, hypochondroplasia, and thanatophoric dysplasia. J Clin Endocrinol Metab. 2015 Feb;100(2):E355-9. doi: 10.1210/jc.2014-2814. Epub 2014 Nov 11. PMID 25387261